CLINICAL TRIAL: NCT00765739
Title: The Effect of Neuromuscular Electrical Stimulation (NMES) in Inducing Muscle Hypertrophy and Improvement in Muscle Torque Output Within the Quadriceps Muscle of Elderly People
Brief Title: The Effect of Neuromuscular Electrical Stimulation (NMES)
Acronym: NMES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMES1
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Muscle Fiber Atrophy, Type II
Keywords: muscle fibers; aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): The group who will get neuromuscular electrical stimulation (NMES)
  Interventions: Other: Neuromuscular electrical stimulation
- 2 (Active Comparator): The group who will do the voluntary muscle contraction
  Interventions: Other: voluntary strengthening exercise

INTERVENTIONS:
Other: Neuromuscular electrical stimulation — neuromuscular electrical stimulation that produce 40% of the maximum voluntary contraction
  Arms: 1
Other: voluntary strengthening exercise — contracting the quadriceps muscle voluntarily to produce 40% of maximum voluntary contraction
  Arms: 2

SUMMARY:
The purpose of this project is to test the effectiveness of neuromuscular electrical stimulation (NMES) that produces 40 % of maximum voluntary contraction (MVC) in increasing muscle size and improvement in muscle force output within the thigh muscle of elderly people.

DETAILED DESCRIPTION:
Declines in whole skeletal muscle strength and size are features commonly associated with aging. Aging reduces the number of fibers in the whole muscle, which explains the loss of muscle mass. Frontera et al studied muscle strength, cross sectional area, and contractile properties of skinned parts of single fibers of the quadriceps muscle. He found that the strength and the whole muscle cross sectional area of knee extensors were significantly higher in young men compared to old subjects, but there were no differences between old and young subjects when the whole muscle strength was adjusted to the whole muscle cross sectional area (specific tension). He also found that muscle fibers from young men were stronger than muscle fibers from old men expressing the same myosin heavy chain isoform even after adjusting for size. Therefore they concluded that abnormality in the quantity and/or function of the contractile or regulatory proteins could explain the reduction in the ability of muscle fibers to generate force.

Along with the loss of muscle fibers, atrophy of the fibers also has been attributed to the aging process. This atrophy has been found to be selective to type II muscle fibers. Lexel et al found in a study done on the cross sections of the whole vastus lateralis muscle from 20 men (19-84 years of age) that the mean Cross Sectional Area (CSA) of type II fibers from muscles of older individuals was on average 35 % smaller while the mean CSA of type I was approximately 6 % smaller than that of young individuals.

Aging and muscles Maintaining muscle strength and size with aging has become a significant issue for elderly trying to keep up independent living and good quality of life. Several studies on old men and women have proven the effectiveness of the resistance exercises in reversing sarcopenia related problems . However in order to increase the size of type II muscle fibers we need to apply high intensity exercises (80 % of 1 RM), or by applying low resistance exercise that is very intense and is done with a large number of repetitions.

The use of electrical stimulation is well documented to improve quadriceps femoris muscle torque output. Numerous experiments have been done to characterize the pattern of activation of muscle fibers during electrically stimulated muscle contraction, and the results show that the recruitment of motor units during electrically induced muscle contraction is non selective. In other words, both type I and II fibers may have equal chance of being recruited during electrically induced muscle contraction. It has been found that NMES is more likely to activate type II muscle fibers at relatively low force levels compared to voluntary exercise. If this is found to be true, then we may have an alternative intervention to improve muscle strength and muscle hypertrophy for elderly individuals who could not perform high intensity exercises to achieve these same benefits. This alternative approach might result in improved overall physical function for these individuals.

The quadriceps muscle has been proposed to be treated because there is significant relationship between quadriceps muscle strength and dynamic stability during chair rise and gait at preferred speed in functionally limited elderly individuals

Methods This study is a two group, repeated measures, randomized clinical trial. Baseline measurements of quadriceps muscle cross-sectional area, type II muscle fiber cross-sectional area, quadriceps power output, the timed up and go test, the SPPB, stair climbing test and ramp up power test will be obtained from subjects prior to the interventions. Following the baseline assessments subjects will be randomly assigned to either the NMES group or the comparable isometric strengthening exercise group. A set of sequentially numbered envelopes will be created and a document indicating the intervention assignment will be placed in the sequentially numbered envelopes. Upon completion of the baseline assessment, the study coordinator will take the next envelope in the sequence and open the envelope. The study coordinator will assign the subject to a group based on the randomized group assignment information obtained from the sealed envelop. During the intervention period of the study subjects will receive either NMES or isometric strengthening exercise 3 times a week for 12 weeks. Each session will last from 15-30 minutes. Post training outcome measures will be taken at the end of the 12 week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* 65-80 years old, are walking independently without assistive devices.

Exclusion Criteria:

* Uncontrolled hypertension (defined as the following: 1) if not taking BP medication and resting systolic BP is greater than 140 or diastolic greater than 90, or 2) if taking BP medication and resting systolic BP greater than 160 or diastolic greater than 100).
* History of cardiovascular disease
* History of neurological disorders that effect lower extremity function (stroke, peripheral neuropathy, Parkinson's disease, multiple sclerosis)
* One cortico-steroid injection to the quadriceps or patellar tendon in the past month or 3 within the past year.
* History of quadriceps tendon rupture, patellar tendon rupture, or patellar fracture, which could place them at risk of re-injury during quadriceps strength testing.
* Current pain in the knee or in the thigh muscles.
* Diagnosis of inflammatory arthritis (Rheumatoid arthritis, gout, or psoriatic arthritis)
* Muscle diseases such as muscular dystrophy.
* Currently been participating in a regular exercise program more than 1x/week.
* Been using anticoagulants and platelet inhibitors
* History of chronic and significant respiratory disease or shortness of breath
* Visual impairments to the extent that they can not accurately see the monitor screen during training program.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Cross sectional area of type II muscle fibers | Base line and 3 months follow up

SECONDARY OUTCOMES:
Quadriceps muscle power output | baseline and 3 month follow up
Functional performance | baseline and 3 month follow up
Quadriceps muscle cross sectional area | baseline and 3 month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health and Rehabilitation Sciences, Pittsburgh, Pennsylvania, United States